CLINICAL TRIAL: NCT01586013
Title: Importance of Age as Covariable in the Requirements to Determine the Drug Plasma -Site Effect Equilibration Time for TCI Propofol Pharmacokinetic Models
Brief Title: the Effect Site Equilibration Time of Propofol is Age Dependant
Acronym: ke0agedep
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad del Desarrollo (Other)
Responsible Party: Principal Investigator, Pablo Sepulveda, Dr Med, Universidad del Desarrollo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PSepulveda_ke0age
Record Dates: First submitted 2012-04-19; First posted 2012-04-26 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: propofol; pharmacodynamic; age; ke0

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- propofol infusion (Experimental): Healthy adults scheduled for elective surgery will receive a computer controlled infusion until obtain the loss of counsiousness (BIS <50). After stoping the infusion we observe the emergency of anesthesia and the correspondant BIS curve. Using the complete loss and recovery curve of BIS we can describe the course of the effect of the drug. Venous sample will be taken during the study to evaluate the pharmacokinetic performance of the model.
  Interventions: Drug: evaluation of propofol effect using BIS

INTERVENTIONS:
Drug: evaluation of propofol effect using BIS — propofol administered in target controlled infusion using the pharmacokinetic model of White
  Other Names: evaluation of effect of intravenous di-isopropilfenol

SUMMARY:
This study obtains an effect site model for White (Modified Marsh) pharmacokinetic propofol model. The plasma effect-site rate constant (ke0) obtained is affected by age.

DETAILED DESCRIPTION:
In the Target Controlled Infusion pumps the first order plasma-effect-site steady-state rate constant (ke0) links the pharmacokinetics (PK) and pharmacodynamics (PD) for a given drug and it is used to predict the course of the effect and to calculate a theoretical drug concentration at the effect site. The PK model for propofol recently published by White et al. (derived from the Marsh model used by the Diprifusor®) include covariate as age and gender to describe the pharmacokinetics but does not incorporate a ke0.

Methods: 45 healthy adult patients will be scheduled for elective surgery with standard monitoring and BIS XP (Aspect) will received a White PK model-driven plasma target controlled infusion of propofol ( 12 ugml-1 or 10 ugml-1 over 65 years) to be reached in 4 min. After reaching the target, the infusion will be stopped obtaining a complete effect curve upon patient awakening. Calculated plasma concentration and EEG data were stored every one second. Loss (LOC) and recovery (ROC) of consciousness were assessed and recorded. The dynamic relationship between propofol Ce and its effect as measured by BIS will be modeled with an inhibitory Emax model using a population PK/PD approach with NONMEM V.

the Study take around 12 min.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2

Exclusion Criteria:

* less than 70% or more than 130% ideal body mass index,
* neurologic disorders,
* pregnancy,
* psychoactive medication intake during last 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
pharmacodynamic model for the White propofol pharmacokinetic | Bispectral index
  Using a propofol target controlled infusion using de White propofol model, we evaluate a complete curve of depression and recovery of the BIS

CONTACTS AND LOCATIONS:
Overall Officials: Pablo O Sepulveda, Dr, Principal Investigator — Clinica Alemana Universidad del Desarrollo
Locations (1):
- Clinica Alemana, Santiago, Chile

REFERENCES:
- [Background] White M, Kenny GN, Schraag S. Use of target controlled infusion to derive age and gender covariates for propofol clearance. Clin Pharmacokinet. 2008;47(2):119-27. doi: 10.2165/00003088-200847020-00005. PMID 18193918